CLINICAL TRIAL: NCT01026610
Title: A Phase IIb, Open, Multinational, Multi-center, Randomised, Comparative, Parallel Study to Assess the Safety and Antiviral Activity of LB80380 Compared to Entecavir 0.5 mg in Chronic Hepatitis B Patients for 48 Weeks With a Planned Analysis of Efficacy and Safety at Week 24 of the Treatment for Selecting Optimal Dose
Brief Title: Safety and Efficacy Study of LB80380 in the Treatment-naive Patients of Chronic Hepatitis B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BVCL007
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic hepatitis B; LB80380; treatment-naive; entecavir
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — ((1-((2-amino-9H-purin-9-yl)methyl)cyclopropyl)oxy)methylphosphonic acid dipivoxyl; entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LB80380 90 mg (Experimental): LB80380 90 mg (90 mg + placebo), once daily oral dose
  Interventions: Drug: LB80380 90 mg
- LB80380 150 mg (Experimental): LB80380 150 mg (60 mg + 90 mg), once daily oral dose
  Interventions: Drug: LB80380 150 mg
- entecavir 0.5 mg (Active Comparator): entecavir 0.5 mg, once daily oral dose
  Interventions: Drug: entecavir 0.5 mg

INTERVENTIONS:
Drug: LB80380 90 mg — LB80380 90 mg + placebo tablets, once daily, for 48 weeks
  Other Names: LB80380
  Arms: LB80380 90 mg
Drug: LB80380 150 mg — LB80380 60 mg + 90 mg tablets, once daily, for 48 weeks
  Other Names: LB80380
  Arms: LB80380 150 mg
Drug: entecavir 0.5 mg — entecavir 0.5 mg tablet, once daily, for 48 weeks
  Other Names: Baraclude
  Arms: entecavir 0.5 mg

SUMMARY:
The purpose of the study is to investigate the safety and the antiviral activity of two doses of LB80380 for 48 weeks in treatment-naive patients with chronic hepatitis B infection compared to entecavir 0.5 mg.

DETAILED DESCRIPTION:
LB80380, an oral prodrug, is a promising candidate nucleotide analogue with antiviral activity against wild-type HBV. LB80380 is undergoing clinical development by LG Life Sciences for use in the treatment of chronic HBV infection.

In this study, the treatment period is 48-week with 24-week of follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Female or male, 18 to 65 years of age, inclusive
* Chronic hepatitis B
* Not treated with anti-viral therapeutics including interferon or pegylated interferons for more than 12 weeks before Screening
* Not treated with anti-viral therapeutics including interferon or pegylated interferons 6 months within Screening
* Compensated chronic hepatitis B
* HBeAg positive or HBeAg negative
* Elevated serum ALT level (1.2-10 X ULN, inclusive)

Exclusion Criteria:

* Co-infection with hepatitis C or D virus (HCV or HDV) or HIV
* Decompensated liver disease
* Creatinine clearance (calculated by Cockroft-Gault formula) less than 50 ml/min
* Screening alpha-fetoprotein (AFP) value greater than or equal to 50 ng/mL, and a follow-up ultrasonography performed prior to baseline shows findings indicative of HCC
* Treatment with immunomodulatory agent or corticosteroids within 6 months prior to study entry.
* Pregnancy or breast-feeding
* Patient is currently abusing alcohol or illicit drugs
* Significant systemic illnesses other than liver diseases
* Presence of other causes of liver disease
* A history of organ transplantation

Presence of anti-HBs at screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2009-08; Primary Completion 2010-11 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Changes in HBV DNA level (log10) from baseline | At Week 24

SECONDARY OUTCOMES:
Proportion of patients with undetectable serum HBV DNA | At Week 24 or Week 48
Proportion of patients with HBeAg seroconversion | At Week 24 or Week 48
Proportion of patients with ALT normalization | At Week 24 or Week 48
Safety assessment during the whole study period | At Week 24 or Week 48

CONTACTS AND LOCATIONS:
Locations (10):
- Queen Mary Hospital, Hong Kong, China
- South Korea (9):
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - Inha University Hospital, Incheon, Inchen
  - Kyungpook National University Hospital, Daegu
  - Pusan National University Yangsan Hospital, Pusan
  - Kangnam Severance Hospital, Yonsei University, Seoul
  - Korea University Medical Center, Seoul
  - Severance Hospital of Yonsei University, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Ulsan University Hospital, Ulsan

REFERENCES:
- [Background] Fung J, Lai CL, Yuen MF. LB80380: a promising new drug for the treatment of chronic hepatitis B. Expert Opin Investig Drugs. 2008 Oct;17(10):1581-8. doi: 10.1517/13543784.17.10.1581. PMID 18808318
- [Background] Yuen MF, Lee SH, Kang HM, Kim CR, Kim J, Ngai V, Lai CL. Pharmacokinetics of LB80331 and LB80317 following oral administration of LB80380, a new antiviral agent for chronic hepatitis B (CHB), in healthy adult subjects, CHB patients, and mice. Antimicrob Agents Chemother. 2009 May;53(5):1779-85. doi: 10.1128/AAC.01290-08. Epub 2009 Feb 17. PMID 19223649